CLINICAL TRIAL: NCT04127903
Title: The First Hospital of Qinhuangdao, Qinhuangdao, Hebei, China.
Brief Title: The Length of the Right Main Stem Bronchus as a Guide to Right-sided Double-lumen Tube Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 2019A123
Record Dates: First submitted 2019-10-13; First posted 2019-10-16 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Therapeutic Procedural Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Length of Right Main Stem Bronchus >=15mm (Experimental)
  Interventions: Other: the Length of Right Main Stem Bronchus
- the Length of Right Main Stem Bronchus <15mm (Experimental)
  Interventions: Other: the Length of Right Main Stem Bronchus

INTERVENTIONS:
Other: the Length of Right Main Stem Bronchus — The distance between the carina and the proximal margin of the right upper lobe orifice on the coronal plane measured by computerised tomography

SUMMARY:
The Length of the Right Main Stem Bronchus Measured by Computerised Tomography as a Guide to Right-sided Double-lumen Tube Use

DETAILED DESCRIPTION:
The double lumen tube (DLT) is the most popular way to isolate the lungs for thoracic surgery. The variable anatomy of the length of the right main stem bronchus seems to be the main reason clinicians are unwilling to use the right-sided DLT (R-DLT). The factors that could compromise the adequate ventilation of the right lung are mostly the variable length of the Right Main Stem Bronchus and the misalignment of the lateral orifice of the right-sided DLT in regard to the right upper lobe bronchus (RULB). The objectives of this study were to validate an alternative method to estimate the length of the Right Main Stem Bronchus by Computerised Tomography as a Guide to Right-sided Double-lumen Tube Use

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing thoracic surgery

Exclusion Criteria:

1. Age>70 or <18 years
2. ASA classifications >III
3. BMI >35kg/m2
4. Modified Mallampati classification ≥III
5. Thoracic surgery within the last one month
6. Severe cardiopulmonary disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
The incidence of Uniblocker displacement | 1 year
The number of adjust the right-sided double-lumen tube to optimum location | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ximing Qi, Study Director — The First Hospital of Qinhuangdao
Locations (1):
- The first hospital of Qinhuangdao, Qinhuangdao, Hebei, China

REFERENCES:
- [Derived] Liu Z, Liu M, Zhao L, Qi X, Yu Y, Liang S, Yang X, Ma Z. Comparison of the accuracy of three methods measured the length of the right main stem bronchus by chest computed tomography as a guide to the use of right sided double-lumen tube. BMC Anesthesiol. 2022 Aug 18;22(1):264. doi: 10.1186/s12871-022-01744-z. PMID 35982403